CLINICAL TRIAL: NCT05388669
Title: A Phase 3, Open-label, Randomized Study of Lazertinib With Subcutaneous Amivantamab Compared With Intravenous Amivantamab in Patients With EGFR-mutated Advanced or Metastatic Non-small Cell Lung Cancer After Progression on Osimertinib and Chemotherapy
Brief Title: A Study of Lazertinib With Subcutaneous Amivantamab Compared With Intravenous Amivantamab in Participants With Epidermal Growth Factor Receptor (EGFR)-Mutated Advanced or Metastatic Non-small Cell Lung Cancer
Acronym: PALOMA-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109211; 61186372NSC3004 (Other: Janssen Research & Development, LLC); 2022-000525-25 (EudraCT Number); 2024-512045-16-00 (Registry Identifier: EUCT number)
Expanded Access: NCT04599712 (Approved for marketing)
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced or Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib; amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Lazertinib with Amivantamab SC-CF (Experimental): Lazertinib 240 milligrams (mg) will be administered orally once daily. Participants will receive amivantamab subcutaneous and co-formulated with recombinant human hyaluronidase (SC-CF), 1600 mg/ 2240 mg depending on the body weight by manual injection. Participants benefiting from study treatment after primary analysis may continue to receive access to study treatment within the study by transferring to the long-term extension (LTE) Phase.
  Interventions: Drug: Lazertinib; Drug: Amivantamab Subcutaneous and Co-Formulated with Recombinant Human Hyaluronidase (SC CF)
- Arm B: Lazertinib with Amivantamab Intravenous (IV) Infusion (Experimental): Lazertinib 240 mg will be administered orally once. Participants will receive amivantamab, 1050 mg or 1400 mg depending on the body weight as an IV infusion. Participants benefiting from study treatment after primary analysis may continue to receive access to study treatment within the study by transferring to the LTE Phase.
  Interventions: Drug: Lazertinib; Drug: Amivantamab Intravenous

INTERVENTIONS:
Drug: Lazertinib — Lazertinib tablets will be administered orally.
  Other Names: JNJ-73841937; YH25448
Drug: Amivantamab Subcutaneous and Co-Formulated with Recombinant Human Hyaluronidase (SC CF) — Amivantamab injection will be administered subcutaneously by manual injection.
  Other Names: JNJ-61186372
  Arms: Arm A: Lazertinib with Amivantamab SC-CF
Drug: Amivantamab Intravenous — Amivantamab will be administered by IV infusion.
  Other Names: JNJ-61186372
  Arms: Arm B: Lazertinib with Amivantamab Intravenous (IV) Infusion

SUMMARY:
The purpose of the study is to simplify amivantamab intravenous administration and to reduce dose times, by assessing a new formulation of amivantamab, amivantamab subcutaneous and co-formulated with recombinant human hyaluronidase (SC-CF), for subcutaneous administration. This formulation has the potential to enhance both the patient and physician experience with amivantamab by providing easier and accelerated administration.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed, advanced or metastatic non-small cell lung cancer (NSCLC), characterized by either epidermal growth factor receptor (EGFR) Exon 19 deletion (Exon 19del) or Exon 21 leucine 858 to arginine substitution (Exon 21 L858R) mutation by an Food and Drug Administration (FDA)-approved or other validated test of either circulating tumor deoxyribonucleic acid (ctDNA) or tumor tissue in a clinical laboratory improvement amendments (CLIA) certified laboratory (sites in the United Started [US]) or an accredited local laboratory (sites outside of the US)
* Have progressed on or after osimertinib (or another approved 3rd generation epidermal growth factor receptor [EGFR] tyrosine kinase inhibitor [TKI]) and platinum-based chemotherapy (irrespective of order). a) The 3rd generation EGFR TKI must have been administered as the first EGFR TKI for metastatic disease or as the second TKI after prior treatment with first- or second-generation EGFR TKI in participants with metastatic EGFR T790M mutation positive NSCLC. b) Participants who decline or are otherwise ineligible for chemotherapy may be enrolled after discussion with the medical monitor. c) Any adjuvant or neoadjuvant treatment, whether with a 3rd generation EGFR TKI or platinum based chemotherapy, would count towards the prior treatment requirement if the participant experienced disease
* Have at least 1 measurable lesion, according to response evaluation criteria in solid tumors (RECIST) version 1.1
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 1
* Any toxicities from prior anticancer therapy must have resolved to common terminology criteria for adverse events (CTCAE) Version 5.0 Grade 1 or baseline level (except for alopecia [any grade], Grade less than or equal to (<=) 2 peripheral neuropathy, and Grade <=2 hypothyroidism stable on hormone replacement)

Exclusion Criteria:

* Participant has received cytotoxic, investigational, or targeted therapies beyond one regimen of platinum-based chemotherapy and EGFR inhibitors
* Participant has received radiotherapy for palliative purposes less than 7 days prior to randomization
* Participant has symptomatic or progressive brain metastases
* Participant has leptomeningeal disease, or participant has spinal cord compression not definitively treated with surgery or radiation
* Participant has uncontrolled tumor-related pain
* Participant has a medical history of interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (187):
- United States (17):
  - City of Hope Duarte, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - City of Hope Long Beach Elm, Long Beach, California
  - National Jewish Health, Denver, Colorado
  - Baptist Lynn Cancer Institute, Boca Raton, Florida
  - Orlando Health, Orlando, Florida
  - University of Kansas, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Astera Cancer Care, East Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Health Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic Westside, Portland, Oregon
  - University of Pennsylvania Division of Hematology Oncology Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Cancer Specialists, Fairfax, Virginia
- Argentina (6):
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas), Buenos Aires
  - Centro Oncológico Korben, Buenos Aires
  - IADT Instituto Argentino de Diagnostico y Tratamiento, CABA
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Sanatorio Allende, Córdoba
  - Clínica Viedma, Viedma
- Australia (6):
  - Cancer Research SA, Adelaide
  - Chris O'Brien Lifehouse, Camperdown
  - Peter MacCallum Cancer Centre, Melbourne
  - St John of God Hospital Murdoch, Murdoch
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Brazil (16):
  - Fundacao Pio XII, Barretos
  - Cetus Oncologia, Belo Horizonte
  - Instituto Cionc de Ensino e Pesquisa S/S, Curitiba
  - Ynova Pesquisa Clinica, Florianópolis
  - Fundacao Sao Francisco Xavier HMC Unidade de Oncologia, Ipatinga
  - UPCO Unidade de Pesquisa Clinica em Oncologia, Pelotas
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Impar Servicos Hospitalares S/A, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Impar Servicos Hospitalares SA Hospital Nove de Julho, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo
  - Onco Star SP Oncologia Ltda, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- China (32):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Chest hospital, Capital medical university, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Jilin cancer hospital, Changchun
  - The First People's Hospital Of Changzhou, Changzhou
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Southwest Hospital, Chongqing
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - Sun Yat-Sen Memorial Hospital Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Huizhou Municipal Central Hospital, Huizhou
  - Huizhou First Hospital, Huizhou
  - Liuzhou people's Hospital, Liuchow
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Shenzhen People s Hospital, Shenzhen
  - Shenzhen university General Hospital, Shenzhen
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xiangyang
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- France (4):
  - CHU Grenoble, La Tronche
  - Institute Coeur Poumon, Lille
  - CHU de Limoges Hopital Dupuytren, Limoges
  - Hopital Nord, Marseille
- Germany (6):
  - Evangelische Lungenklinik Berlin, Berlin
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg, Georgsmarienhütte
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Munster University Hospital, Münster
  - Oncologianova GmbH, Recklinghausen
  - Onkologische Schwerpunktpraxis, Weinsberg
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (9):
  - Oncologia Medica - Irccs - Istituto Tumori Giovanni Paolo II, Bari
  - A O U Sant Orsola Malpighi, Bologna
  - European Institute of Oncology, Milan
  - Aou San Luigi Gonzaga, Orbassano
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Ospedale S. Maria Delle Croci, Ravenna
  - A.O. San Camillo Forlanini, Roma
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Istituto Clinico Humanitas, Rozzano
- Japan (18):
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Himeji Medical Center, Himeji
  - Kansai Medical University Hospital, Hirakata
  - Kanagawa Cancer Center, Kanagawa
  - Kurashiki Central Hospital, Kurashiki
  - Kurume University Hospital, Kurume
  - Matsusaka Municipal Hospital, Matsusaka
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Hokkaido University Hospital, Sapporo
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Fujita Health University Hospital, Toyoake
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka-shi
  - Wakayama Medical University Hospital, Wakayama
  - National Hospital Organization Iwakuni Clinical Center, Yamaguchi
  - National Hospital Organization Yamaguchi Ube Medical Center, Yamaguchi
- Malaysia (6):
  - Prince Court Medical Centre, Kuala Lumpur
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Beacon Hospital Sdn Bhd, Petaling Jaya
  - Sunway Medical Centre, Petaling Jaya
- Poland (5):
  - Centrum Onkologii im Prof F Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Krakowski Szpital Specjalityczny im. Jana Pawla II, Krakow
  - Mazowieckie Centrum Leczenia Chorob Pluc, Otwock
  - Private Specialist Hospitals - MedPolonia, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Portugal (4):
  - Hospital de Braga, Braga
  - Hospital da Luz, SA, Lisbon
  - Hosp. Cuf Descobertas, Lisbon
  - Ulsm - Hosp. Pedro Hispano, Senhora da Hora
- South Korea (9):
  - National Cancer Center, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - GyeongSang National University Hospital, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (16):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hosp. Univ. Lucus Augusti, Lugo
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. Central de Asturias, Oviedo
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Chang Kung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (3):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
- Turkey (Türkiye) (11):
  - Adana City Hospital, Adana
  - Adana Baskent Hospital, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Gazi University Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Acıbadem Maslak Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - IEU Medical Point Hospital, Izmir
  - Medical Park Samsun Hastanesi, Samsun
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Imperial College Healthcare, London
  - Newcastle Freeman Hospital, Newcastle upon Tyne
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Leighl NB, Akamatsu H, Lim SM, Cheng Y, Minchom AR, Marmarelis ME, Sanborn RE, Chih-Hsin Yang J, Liu B, John T, Massuti B, Spira AI, Lee SH, Wang J, Li J, Liu C, Novello S, Kondo M, Tamiya M, Korbenfeld E, Moskovitz M, Han JY, Alexander M, Joshi R, Felip E, Voon PJ, Danchaivijitr P, Hsu PC, Silva Melo Cruz FJ, Wehler T, Greillier L, Teixeira E, Nguyen D, Sabari JK, Qin A, Kowalski D, Sendur MAN, Xie J, Ghosh D, Alhadab A, Haddish-Berhane N, Clemens PL, Lorenzini P, Verheijen RB, Gamil M, Bauml JM, Baig M, Passaro A; PALOMA-3 Investigators. Subcutaneous Versus Intravenous Amivantamab, Both in Combination With Lazertinib, in Refractory Epidermal Growth Factor Receptor-Mutated Non-Small Cell Lung Cancer: Primary Results From the Phase III PALOMA-3 Study. J Clin Oncol. 2024 Oct 20;42(30):3593-3605. doi: 10.1200/JCO.24.01001. Epub 2024 Jun 10. PMID 38857463

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results are currently reported for primary analysis till clinical cut-off date 03-Jan-2024. Upon completion of the open-label follow-up phase, participants were permitted to enter the long-term extension (LTE) phase. The LTE phase is ongoing and results will be published after the completion of the study.
Groups:
- Arm A: Lazertinib With Amivantamab SC-CF: Participants were administered lazertinib 240 milligrams (mg) tablet orally once daily from Cycle 1 Day 1 until Cycle 15, with each cycle consisting of 28 days. Participants then received amivantamab subcutaneous injection with at dose 1600 mg (if body weight [BW] is less than [<] 80 kilograms [kg]) or 2240 mg (if BW is greater than or equal to [>=] 80 kg) co-formulated (SC-CF) with recombinant human hyaluronidase PH20 (rHuPH20) 160 milligrams per milliliter (mg/mL) through manual injection on Cycle 1 Days 1, 8, 15, and 22, and on Days 1 and 15 of each subsequent cycle, starting from Cycle 2. After the completion of primary analysis, participants who benefited from the study treatment continued their treatment within the study upon transitioning into the LTE phase.
- Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion: Participants were administered lazertinib 240 mg orally once daily from Cycle 1 Day 1 until Cycle 15, with each cycle consisting of 28 days. Participants then received amivantamab intravenous infusion at dose 1050 mg (if BW< 80 kg) or 1400 mg (if BW >=80 kg) on Cycle 1 Days 1-2 (split dose), 8, 15, 22, and on Days 1 and 15 of each subsequent cycle, starting from Cycle 2. After the completion of primary analysis, participants who benefited from the study treatment continued their treatment within the study upon transitioning into the LTE phase.
Period: Overall Study
Arm/Group | Arm A: Lazertinib With Amivantamab SC-CF | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion
Started | 206 | 212
Treated (Safety Analysis) | 206 | 210
Completed | 43 | 62
Not Completed | 163 | 150
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other-Ongoing | 156 | 141

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Lazertinib With Amivantamab SC-CF | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion | Total
Number analyzed (Participants) | 206 | 212 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.76) | 61.4 (10.71) | 61.1 (10.25)
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 28 | 29 | 57
  50-64 years | 105 | 91 | 196
  65-74 years | 55 | 70 | 125
  >=75 years | 18 | 22 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 141 | 279
  Male | 68 | 71 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 126 | 129 | 255
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 78 | 77 | 155
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 5 | 6 | 11
  Australia | 12 | 5 | 17
  Brazil | 6 | 11 | 17
  Canada | 7 | 11 | 18
  China | 46 | 47 | 93
  France | 3 | 4 | 7
  Germany | 2 | 3 | 5
  Israel | 9 | 4 | 13
  Italy | 13 | 14 | 27
  Japan | 26 | 30 | 56
  Malaysia | 8 | 9 | 17
  Poland | 3 | 0 | 3
  Portugal | 3 | 2 | 5
  Korea, South | 21 | 20 | 41
  Spain | 14 | 15 | 29
  Taiwan | 6 | 6 | 12
  Thailand | 5 | 2 | 7
  Turkey | 5 | 2 | 7
  United Kingdom | 0 | 2 | 2
  United States | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: For All Regions Other Than the European Union (EU) and Others Accepting Cycle 2 Day 1: Observed Serum Concentration (Ctrough) of Amivantamab at Steady State
Description: Ctrough was the observed serum concentration of Amivantamab at steady state immediately prior to the next drug administration.
Time Frame: Pre-dose on Cycle 4 Day 1 (each cycle of 28 days)
Population: The pharmacokinetic (PK) primary endpoint evaluable set included all randomized participants who had received all doses in Cycle 1-3, without dose modifications and provided Cycle 4 Day 1 Ctrough. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (mcg/mL)
Arm/Group | Arm A: Lazertinib With Amivantamab SC-CF | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion
Number analyzed (Participants) | 98 | 98
micrograms per milliliters (mcg/mL) | 206 (39.1) | 144 (41.5)
Statistical Analysis 1: Comparison: Arm A: Lazertinib With Amivantamab SC-CF vs Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion; Arm B Vs Arm A; Test type: Non-Inferiority — The primary hypothesis tests was based on one-sided test at significance level of alpha = 0.05 to demonstrate the non-inferiority of the amivantamab SC-CF relative to amivantamab IV; Cox regression model = 1.427, 90% CI 2-sided [1.266 to 1.610]

2. Primary Outcome: For EU and Any Applicable Region: Observed Serum Concentration (Ctrough) of Amivantamab
Description: Ctrough was the observed serum concentration of Amivantamab immediately prior to the next drug administration.
Time Frame: Pre-dose on Cycle 2 Day 1 (each cycle of 28 days)
Population: The PK primary endpoint evaluable set included all randomized participants who had received all doses in Cycle 1, without dose modifications and provided Cycle 2 Day 1 Ctrough. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Arm A: Lazertinib With Amivantamab SC-CF | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion
Number analyzed (Participants) | 160 | 142
mcg/mL | 335 (32.7) | 293 (31.7)
Statistical Analysis 1: Comparison: Arm A: Lazertinib With Amivantamab SC-CF vs Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion; Arm B Vs Arm A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Cox regression model = 1.145, 90% CI 2-sided [1.040 to 1.261]

3. Primary Outcome: Area Under the Concentration (AUC) Time Curve of Amivantamab From Day 1 to Day 15 (AUC [Day 1-15]) of Cycle 2
Description: AUC (Day 1-15) defined as area under the concentration time curve from Cycle 2 Day 1 to Day 15 were reported.
Time Frame: Cycle 2: Arm A: pre-dose, 24, 48, 72, 96, 168, and 360 hours (hrs) post-dose on Day 1; Arm B: pre-infusion, end of infusion (EOI)+10 minutes, EOI+2, EOI+6, EOI+24, EOI+48, EOI+72, EOI+168, and EOI+360 hrs post dose on Day 1
Population: The PK primary endpoint evaluable set included all randomized participants who had received all doses up to Cycle 2 Day 1, without dose modifications and provided all necessary PK samples to derive primary PK endpoint Cycle 2 AUC(D1-D15). Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliters
Arm/Group | Arm A: Lazertinib With Amivantamab SC-CF | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion
Number analyzed (Participants) | 140 | 132
micrograms*hour per milliliters | 135861 (30.7) | 131704 (24.0)
Statistical Analysis 1: Comparison: Arm A: Lazertinib With Amivantamab SC-CF vs Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion; Arm B Vs Arm A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.032, 90% CI 2-sided [0.976 to 1.090]

4. Secondary Outcome: Objective Response Rate (ORR)
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Progression-Free Survival (PFS)
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Duration of Response (DOR)
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Time to Response (TTR)
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Number of Participants With AEs by Severity
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

11. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities by Severity
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

12. Secondary Outcome: Number of Participants With Infusion Related Reactions (IRRs)
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

13. Secondary Outcome: Number of Participants With IRRs by Severity
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

14. Secondary Outcome: For All Regions Other Than the EU and Others Accepting Cycle 2 Day 1: Observed Serum Concentration (Ctrough) of Amivantamab at Pre-dose on Cycle 2 Day 1
Time Frame: Pre-dose on Cycle 2 Day 1 (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2026-12

15. Secondary Outcome: For EU and Any Applicable Region: Observed Serum Concentration (Ctrough) of Amivantamab at Steady State on Cycle 4 Day 1
Time Frame: Pre-dose on Cycle 4 Day 1 (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2026-12

16. Secondary Outcome: Model-Predicted Area Under the Concentration Time Curve of Amivantamab at Steady State From Day 1 to Day 15 (AUC [Day 1-15]) of Cycle 4
Time Frame: Cycle 4: Arm A: pre-dose, 24, 48, 72, 96, 168, and 360 hrs post-dose on Day 1; Arm B: preinfusion, EOI+10 minutes, EOI+2, EOI+6, EOI+24, EOI+48, EOI+72, EOI+168, and EOI+360 hrs post dose on Day 1
Reporting Status: Not Posted, anticipated posting 2026-12

17. Secondary Outcome: Percentage of Participants With Presence of Anti-amivantamab Antibodies and Anti-rHuPH20 Antibodies
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

18. Secondary Outcome: Percentage of Participants With Cancer Therapy Satisfaction as Assessed by Therapy Administration Satisfaction Questionnaire (TASQ)
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

19. Secondary Outcome: Change From Baseline in Therapy Administration Satisfaction Questionnaire (TASQ) as Assessed Over Time
Time Frame: From baseline (Day 1, Cycle 1) to 3 years 4 months (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2026-12

20. Secondary Outcome: Participant Chair Time
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

21. Secondary Outcome: Participant Chair Time in Treatment Room
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

22. Secondary Outcome: Duration of Treatment Administration
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

23. Secondary Outcome: Active Health Care Professional (HCP) Time For Drug Preparation, Treatment Administration and Post-treatment Monitoring
Time Frame: Up to 3 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: All cause mortality: From baseline (Day 1) up to 17 months; SAEs and other AEs: From baseline (Day 1) up to 8 months
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Arm A: Lazertinib With Amivantamab SC-CF | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion
All-Cause Mortality (participants affected / at risk) | 43/206 | 61/210
Serious Adverse Events (participants affected / at risk) | 59/206 | 64/210
Other Adverse Events (participants affected / at risk) | 201/206 | 207/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Lazertinib With Amivantamab SC-CF (N=206) | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion (N=210)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Oesophageal Stenosis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 2
Fatigue (General disorders) | 3 | 1
Pyrexia (General disorders) | 1 | 1
Sudden Death (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Bacterial Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 4 | 4
Herpes Simplex (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Myiasis (Infections and infestations) | 1 | 0
Oral Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 7
Pneumonia Aspiration (Infections and infestations) | 0 | 1
Pneumonia Viral (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 2
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 4 | 3
Aspartate Aminotransferase Increased (Investigations) | 1 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 3
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Capillary Leak Syndrome (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 2 | 4
Embolism Arterial (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Lazertinib With Amivantamab SC-CF (N=206) | Arm B: Lazertinib With Amivantamab Intravenous (IV) Infusion (N=210)
Anaemia (Blood and lymphatic system disorders) | 39 | 40
Leukopenia (Blood and lymphatic system disorders) | 12 | 8
Lymphopenia (Blood and lymphatic system disorders) | 8 | 19
Neutropenia (Blood and lymphatic system disorders) | 12 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 29 | 33
Constipation (Gastrointestinal disorders) | 42 | 42
Diarrhoea (Gastrointestinal disorders) | 43 | 39
Gingival Bleeding (Gastrointestinal disorders) | 16 | 13
Haemorrhoids (Gastrointestinal disorders) | 12 | 6
Nausea (Gastrointestinal disorders) | 60 | 52
Stomatitis (Gastrointestinal disorders) | 57 | 69
Vomiting (Gastrointestinal disorders) | 43 | 41
Asthenia (General disorders) | 31 | 21
Fatigue (General disorders) | 43 | 42
Malaise (General disorders) | 17 | 11
Oedema Peripheral (General disorders) | 52 | 58
Pyrexia (General disorders) | 24 | 20
Hyperbilirubinaemia (Hepatobiliary disorders) | 15 | 6
Conjunctivitis (Infections and infestations) | 14 | 10
Covid-19 (Infections and infestations) | 13 | 15
Paronychia (Infections and infestations) | 111 | 108
Urinary Tract Infection (Infections and infestations) | 4 | 11
Administration Related Reaction (Injury, poisoning and procedural complications) | 20 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 27 | 137
Alanine Aminotransferase Increased (Investigations) | 46 | 54
Aspartate Aminotransferase Increased (Investigations) | 42 | 44
Blood Alkaline Phosphatase Increased (Investigations) | 22 | 20
Blood Creatinine Increased (Investigations) | 15 | 14
Blood Lactate Dehydrogenase Increased (Investigations) | 19 | 13
Gamma-Glutamyltransferase Increased (Investigations) | 21 | 14
Weight Decreased (Investigations) | 25 | 15
Decreased Appetite (Metabolism and nutrition disorders) | 45 | 52
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 96 | 76
Hypocalcaemia (Metabolism and nutrition disorders) | 33 | 27
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 19
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 17 | 22
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 17 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 13
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 26 | 20
Dizziness (Nervous system disorders) | 23 | 24
Headache (Nervous system disorders) | 42 | 36
Hypoaesthesia (Nervous system disorders) | 8 | 11
Peripheral Sensory Neuropathy (Nervous system disorders) | 16 | 19
Insomnia (Psychiatric disorders) | 15 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 15
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 64 | 69
Dry Skin (Skin and subcutaneous tissue disorders) | 24 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 25
Rash (Skin and subcutaneous tissue disorders) | 95 | 91
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 11 | 10
Skin Fissures (Skin and subcutaneous tissue disorders) | 15 | 15
Hypotension (Vascular disorders) | 6 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT05388669/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT05388669/SAP_001.pdf